CLINICAL TRIAL: NCT07085468
Title: A Parallel-Group, Double-Blind Study to Investigate the Safety and Tolerability of LY3549492 Compared With Placebo in Adult Participants Aged 55 to 80 Years With a BMI of 22 to 25 kg/m2
Brief Title: A Study of LY3549492 in Healthy Weight Adult Participants
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated for strategic business reasons
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 27357; J3H-MC-GZNI (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Elderly; Body Weight; Body Composition
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3549492 Dose 1 (Experimental): Participants will receive LY3549492 orally
  Interventions: Drug: LY3549492
- LY3549492 Dose 2 (Experimental): Participants will receive LY3549492 orally
  Interventions: Drug: LY3549492
- Placebo (Placebo Comparator): Participants will receive placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3549492 — Administered orally
  Arms: LY3549492 Dose 1; LY3549492 Dose 2
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3549492 in adult participants with a healthy body max index (BMI) of 22 to 25 kilograms per square meter (kg/m2).

Participation in the study will last about 13 months.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) within the range of 22 to 25 kilograms per square meter (kg/m2)
* Have had a stable body weight for 3 months prior to screening

Exclusion Criteria:

* Have type 1 diabetes, latent autoimmune diabetes in adults, or a history of ketoacidosis or hyperosmolar coma
* Have:

  * type 2 diabetes and on antidiabetic therapy (except type 2 diabetes being managed with diet and/or stable dose of metformin)
  * rare forms of diabetes mellitus, or
  * hemoglobin A1c (HbA1c) >8%
* Have poorly controlled hypertension
* Have any of the following cardiovascular conditions within 12 months prior to screening:

  * acute myocardial infarction
  * stroke
  * unstable angina, or
  * hospitalization due to congestive heart failure.
* Have a history of New York Heart Association Functional Classification III or IV congestive heart failure
* Have signs and symptoms of liver disease
* Have a history of pancreatitis
* Have taken medications or alternative remedies for weight loss or weight gain within 3 months prior to screening

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-07-21 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Events (SAE) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Week 48
  A summary of treatment emergent adverse events (TEAEs), SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module.

SECONDARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 24, Week 48
Number of Participants with Adverse Events Leading to Permanent Discontinuation of Study Intervention or Withdrawal | Baseline through Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- United States (11):
  - Headlands Research - Scottsdale, Scottsdale, Arizona
  - Valley Clinical Trials, Inc., Covina, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Artemis Institute for Clinical Research, San Diego, California
  - JEM Research Institute, Atlantis, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Great Lakes Clinical Trials - Andersonville, Chicago, Illinois
  - Alliance for Multispecialty Research, LLC, Lexington, Kentucky
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - Trial Management Associates, Myrtle Beach, South Carolina
- Canada (10):
  - Viacar Recherche Clinique, Greenfield Park
  - Apex Trials, Guelph
  - OCT Research ULC, Kelowna
  - Clinique Mémoire de Montréal, Montreal
  - Ottawa Memory Clinic, Ottawa
  - Richmond Clinical Trials, Richmond
  - Q&T Research Sherbrooke Inc., Sherbrooke
  - Toronto Memory Program, Toronto
  - BioPharma Services, Toronto
  - Diex Recherche Trois-Rivieres, Trois-Rivières

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/